CLINICAL TRIAL: NCT00684138
Title: ACRYSOF® ReSTOR® Aspheric +3.0 D Add Power Intraocular Lens (IOL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Tonya Tubbs Jones, Alcon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-06-40
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Cataract
Keywords: cataract; cataract surgery; IOL; intraocular lens; ReSTOR; Replacement of cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReSTOR Aspheric +3.0D (Experimental): ACRYSOF® ReSTOR® Aspheric +3.0 D Add Power Intraocular Lens
  Interventions: Device: ACRYSOF® ReSTOR® Aspheric +3.0 D Add Power Intraocular Lens
- ReSTOR Aspheric +4.0D (Active Comparator): ACRYSOF® ReSTOR® Aspheric +4.0 D Add Power Intraocular Lens
  Interventions: Device: ACRYSOF® ReSTOR® Aspheric +4.0 D Add Power Intraocular Lens

INTERVENTIONS:
Device: ACRYSOF® ReSTOR® Aspheric +4.0 D Add Power Intraocular Lens — Intraocular Lens
  Arms: ReSTOR Aspheric +4.0D
Device: ACRYSOF® ReSTOR® Aspheric +3.0 D Add Power Intraocular Lens — Intraocular Lens
  Arms: ReSTOR Aspheric +3.0D

SUMMARY:
Randomized, parallel group, subject masked, multi-center six (6) month follow-up study comparing ACRYSOF® ReSTOR® Aspheric +3.0 D Add Power IOL Model SN6AD1 implanted in both eyes to ACRYSOF® ReSTOR® Aspheric +4.0 D Add Power IOL Model SN6AD3 implanted in both eyes.

ELIGIBILITY:
Inclusion:

* Adults, 21 years of age or older at the time of surgery, of either gender or any race, diagnosed with bilateral cataracts
* Calculated lens power is within the available range
* Willing and able to complete all required postoperative visits
* Planned cataract removal by phacoemulsification and/or liquifacture
* Potential postoperative visual acuity of 0.2 logMAR or better in study eyes
* Preoperative astigmatism of 1.0 Diopter (D) or less, measured by keratometry in study eyes
* Clear intraocular media other than cataract in study eyes
* Able to comprehend and sign a statement of informed consent
* Preoperative Best Corrected Distance Visual Acuity (BCDVA) worse than 0.2 logMAR, or if BCDVA is equal to or better than 0.2 logMAR, BCDVA with a Brightness Acuity Tester (BAT) on "Medium" setting must be worse than 0.2 logMAR

Exclusion:

* Significant irregular corneal aberration as demonstrated by corneal topography
* Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause future acuity losses to a level worse than 0.2 logMAR
* Subjects who may reasonably be expected to require laser treatments at any time
* Previous corneal refractive surgery
* Amblyopia
* Clinically severe corneal dystrophy (e.g., epithelial, stromal, or endothelial dystrophy)
* Diabetic retinopathy
* Extremely shallow anterior chamber, not due to swollen cataract
* Microphthalmos
* Previous retinal detachment
* Previous corneal transplant
* Recurrent severe anterior or posterior segment inflammation of unknown etiology
* Rubella or traumatic cataract
* Iris neovascularization
* Glaucoma (uncontrolled or controlled with medication)
* Aniridia
* Optic nerve atrophy
* Pregnancy
* Current or previous usage of an alpha-1-selective adrenoceptor blocking agent or an antagonist of alpha 1A adrenoceptor (e.g.Flomax® (tamsulosin HCL), Hytrin®, or Cardura®)
* Any subject currently participating in another investigational drug or device study that may confound the results of this investigation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Call Center for Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only adult subjects of either gender or any race in need of cataract extraction in both eyes were considered for enrollment. 280 subjects were implanted bilaterally with either the ACRYSOF® ReSTOR® Aspheric +3.0 D Add Power IOL Model SN6AD1 or the ACRYSOF® ReSTOR® Aspheric +4.0 D Add Power IOL Model SN6AD3 based upon a 1:1 randomization.
Pre-assignment Details: Subjects were examined to ensure inclusion/exclusion criteria. Only subjects who signed an informed consent and qualified to be in the study were enrolled. Subject numbers were assigned after obtaining consent meeting inclusion/exclusion criteria. Subjects were considered enrolled once implanted in the first operative eye.
Groups:
- ACRYSOF® ReSTOR® +3.0: ACRYSOF® ReSTOR® Aspheric +3.0 D Add Power Intraocular Lens
- ACRYSOF® ReSTOR® Aspheric +4.0: ACRYSOF® ReSTOR® Aspheric +4.0 D Add Power Intraocular Lens
Period: Overall Study
Arm/Group | ACRYSOF® ReSTOR® +3.0 | ACRYSOF® ReSTOR® Aspheric +4.0
Started | 141 | 139
Completed | 138 | 131
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACRYSOF® ReSTOR® +3.0 | ACRYSOF® ReSTOR® Aspheric +4.0 | Total
Number analyzed (Participants) | 141 | 139 | 280
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 40 | 91
  >=65 years | 90 | 99 | 189
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 97 | 192
  Male | 46 | 42 | 88

OUTCOME MEASURES:

1. Primary Outcome: Binocular Distance Corrected Near Visual Acuity at Best Distance (That Which Provides the Subject With the Best Vision)
Description: Binocular Distance Corrected Near Visual Acuity at Best Distance (that which provides the subject with the best vision)measured in mean logMAR. logMAR is the logarithm of the minimum angle of resolution, which is a measure for visual acuity (VA). Mean logMAR is the average value of visual acuity.
Time Frame: 3 months
Population: Only patients bilaterally implanted with the test article were considered for the outcome measures. One study lens was removed following implantation, but prior to surgery completion, resulting in 279 subjects who were implanted and available for postoperative follow-up (evaluable for All Implanted Analysis).
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | ACRYSOF® ReSTOR® +3.0 | ACRYSOF® ReSTOR® Aspheric +4.0
Number analyzed (Participants) | 138 | 131
logMAR | 0.07 [0.0539 to 0.0854] | 0.09 [0.0854 to 0.1081]

2. Secondary Outcome: Binocular Distance Corrected Distance Visual Acuity
Description: Binocular Distance Corrected Distance Visual Acuity measured in logMAR. LogMAR is the logarithm of the minimum angle of resolution, which is a measure for visual acuity (VA).
Time Frame: 3 months post-operative
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | ACRYSOF® ReSTOR® +3.0 | ACRYSOF® ReSTOR® Aspheric +4.0
Number analyzed (Participants) | 138 | 131
logMAR | -0.05 [-0.065 to -0.040] | -0.05 [-0.061 to -0.039]

3. Secondary Outcome: Binocular Distance Corrected Intermediate Visual Acuity (Tested at 50 cm)
Description: Binocular Distance Corrected Intermediate Visual Acuity (tested at 50 cm) measured in logMAR. LogMAR is the logarithm of the minimum angle of resolution, which is a measure for visual acuity (VA).
Time Frame: 3 months post-operative
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | ACRYSOF® ReSTOR® +3.0 | ACRYSOF® ReSTOR® Aspheric +4.0
Number analyzed (Participants) | 138 | 131
logMAR | 0.06 [0.0384 to 0.0849] | 0.24 [0.2188 to 0.2667]

4. Secondary Outcome: Binocular Distance Corrected Intermediate Visual Acuity (Tested at 60 cm)
Description: Binocular Distance Corrected Intermediate Visual Acuity (tested at 60 cm)measured in logMAR. LogMAR is the logarithm of the minimum angle of resolution, which is a measure for visual acuity (VA).
Time Frame: 3 months post-operative
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | ACRYSOF® ReSTOR® +3.0 | ACRYSOF® ReSTOR® Aspheric +4.0
Number analyzed (Participants) | 138 | 131
logMAR | 0.12 [0.0916 to 0.1381] | 0.32 [0.2972 to 0.3451]

5. Secondary Outcome: Binocular Distance Corrected Intermediate Visual Acuity (Tested at 70 cm)
Description: Binocular Distance Corrected Intermediate Visual Acuity (tested at 70 cm) measured in logMAR. LogMAR is the logarithm of the minimum angle of resolution, which is a measure for visual acuity (VA).
Time Frame: 3 months post-operative
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | ACRYSOF® ReSTOR® +3.0 | ACRYSOF® ReSTOR® Aspheric +4.0
Number analyzed (Participants) | 138 | 131
logMAR | 0.18 [0.1597 to 0.2062] | 0.34 [0.3190 to 0.3669]

ADVERSE EVENTS:
Time Frame: Up to six months after cataract surgery.
Description: Adverse events were collected from the time of cataract surgery until pre-market approval submission for all 300 patients enrolled in the study.
Groups:
- ACRYSOF® ReSTOR® +3.0 (First Eyes): ACRYSOF® ReSTOR® Aspheric +3.0 D Add Power Intraocular Lens - First eye implanted only
- ACRYSOF® ReSTOR® Aspheric +4.0 (First Eyes): ACRYSOF® ReSTOR® Aspheric +4.0 D Add Power Intraocular Lens - First eye implanted only
- ACRYSOF® ReSTOR® +3.0 (Second Eyes): ACRYSOF® ReSTOR® Aspheric +3.0 D Add Power Intraocular Lens - Second eye implanted only
- ACRYSOF® ReSTOR® Aspheric +4.0 (Second Eyes): ACRYSOF® ReSTOR® Aspheric +4.0 D Add Power Intraocular Lens - Second eye implanted only
Arm/Group | ACRYSOF® ReSTOR® +3.0 (First Eyes) | ACRYSOF® ReSTOR® Aspheric +4.0 (First Eyes) | ACRYSOF® ReSTOR® +3.0 (Second Eyes) | ACRYSOF® ReSTOR® Aspheric +4.0 (Second Eyes)
Serious Adverse Events (participants affected / at risk) | 6/153 | 2/147 | 2/151 | 3/143
Other Adverse Events (participants affected / at risk) | 0/153 | 0/147 | 0/151 | 0/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACRYSOF® ReSTOR® +3.0 (First Eyes) (N=153) | ACRYSOF® ReSTOR® Aspheric +4.0 (First Eyes) (N=147) | ACRYSOF® ReSTOR® +3.0 (Second Eyes) (N=151) | ACRYSOF® ReSTOR® Aspheric +4.0 (Second Eyes) (N=143)
Hypopyon (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endophthalmitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular Edema (Eye disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Lens Dislocation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical reintervention (SI) (Surgical and medical procedures) | 2 (5) | 1 (1) | 2 (2) | 2 (2) — Some eyes experienced SI and more than 1 SAE. SN5AD1 (1st Eye): 1 patient - hypopyon, endophthalmitis; 1 patient - lens dislocation; and 1 patient - after the close of the study. SN6AD3 (1st Eye): 1 patient - later had macular edema.

LIMITATIONS AND CAVEATS:
Data from one investigator, who implanted 20 subjects, were excluded from analysis due to non compliance with data collection and documentation. This resulted in 280 implanted subjects that were considered evaluable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other